CLINICAL TRIAL: NCT02556840
Title: Impact of Two Standardized Clinical Care Protocols on Pregnancy Outcomes in Women With Monogenic Diabetes MODY2
Brief Title: Impact on Birth Weight of Two Therapeutic Strategies (Insulin Therapy From the Beginning of Pregnancy vs. Insulin Therapy Initiated According to Fetal Growth Evaluated by Ultrasonography Measurements) in Pregnant Women With Monogenic Diabetes
Acronym: MODY2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-A00261-48
Record Dates: First submitted 2015-07-13; First posted 2015-09-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Maturity-Onset Diabetes of the Young
Keywords: Monogenic diabetes; maturity-onset diabetes of the young; MODY; Pregnancy; Gestational diabetes; Glucokinase; Insulin therapy during pregnancy; Evaluation of fetal growth by ultrasonography measurements
MeSH Terms: conditions — Mason-Type Diabetes; Diabetes Mellitus, Type 2; Diabetes, Gestational; Maturity-Onset Diabetes of the Young, Type 2 | interventions — Convulsive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin therapy from the beginning of pregnancy (Active Comparator): Insulin therapy (Glargine/Lantus®, Détémir/Levemir® , Insulatard® , Umuline NPH® , Lispro/Humalog® , Asparte/Novorapid® or Actrapid ®) administered from the beginning of pregnancy according to maternal blood glucose (if fasting blood glucose > 0.95g/l or post-prandial blood glucose > 1.20g/l) as recommended by the national guidelines for gestational diabetes mellitus.
  Insulin administered to patients either by subcutaneous injections or by pump.
  Interventions: Other: insulin therapy
- Insulin therapy initiated according to fetal growth (Experimental): Insulin therapy (Glargine/Lantus®, Détémir/Levemir® , Insulatard® , Umuline NPH® , Lispro/Humalog® , Asparte/Novorapid® or Actrapid ®) initiated according to fetal growth evaluated by ultrasonography measurements. MODY2 women will not be treated with insulin until delivery, except when the fetal abdominal circumference exceeds ≥ the 75 percentile on one US or maternal fasting capillary blood glucose is ≥ 1,20 g/L or maternal post-prandial capillary blood glucose is ≥ 2,00 g/L.
  Insulin administered to patients either by subcutaneous injections or by pump.
  Interventions: Other: insulin therapy

INTERVENTIONS:
Other: insulin therapy

SUMMARY:
Maturity-onset diabetes of youth (MODY) are the most frequent monogenic diabetes with autosomic dominant inheritance (2% of diabetes). The MODY2 diabetes is related to a defect in the glucokinase (GCK) enzyme, the first limiting step of insulin secretion. An abnormal GCK leads to a delayed insulin secretion. Patients with GCK mutations have only mild raised fasting plasma glucose. Treatment is usually unnecessary since hyperglycemia is stable and MODY2 patients have no microvascular complications of diabetes. In contrast, pregnancy in MODY2 women is a challenging situation. A non-mutated fetus will produce excess insulin in response to raised maternal blood glucose leading to an accelerated growth and a higher risk of macrosomia. The mother of non-mutated fetus should therefore be treated to normalize her blood glucose levels. On contrary, a mutated fetus will produce a delayed insulin secretion (as his MODY2 mother) in response to maternal hyperglycemia. Consequently insulin therapy during pregnancy would reduce fetal insulin secretion and result in a low birth weight.

Moreover, insulin therapy exposes pregnant women to more labor induction, prematurity and cesarean deliveries. In these MODY2 women whose glucose set point is physiologically higher, glycemic goals are difficult to achieve while often requiring extensive insulin therapy. An optimal situation would consist in initiating insulin therapy only for women with non-mutated offsprings. Unfortunately no antenatal diagnosis of the GCK mutation on fetal cells is available yet. In literature, birth weight differences between mutated and non-mutated neonates may reach up to 700g. In clinical practice, two strategies are used but without standardized protocol on glycemic targets, delay and doses of insulin : 1) insulin at diagnosis of pregnancy 2) treatment based on fetal abdominal circumference and fetal weight measurements by ultrasonography (US) and initiated if fetal biometry is greater than the 75th percentile.

The purpose of the study is to evaluate for the first time these two management strategies through a prospective and standardized study. Hypothesis: US assessment would be sufficient to identify fetuses at risk of macrosomia and to initiate insulin treatment in mothers.

DETAILED DESCRIPTION:
Study design The investigators propose to conduct a national multicenter prospective study on the clinical management of pregnancy in women with GCK mutations.

Medical management of the pregnancy After obtaining written informed consent, each investigator of the Diabetes Departments will include MODY2 women, at the time of gestation planning or at the first prenatal appointment. Pre-gestational maternal parameters (maternal age, pre-gestational weight, blood glucose, mean blood glucose levels before and 2 hours post prandial over one week when available, HbA1c, parity, medical history of macrosomia) will be collected.

Antenatal care will be provided according to the local routine protocol for MODY2. All women will receive dietary and physical activity counselling according to current recommendations for pregnant women with pregestational diabetes. Vitamin B9, 0.4 or 5 mg/day, according to local habits, will be prescribed as usual care from pregestational appointment until the end of first trimester.

* Women with a pregestational HbA1c ≥ 6.5 % will be systematically treated with insulin because of a potential increase in the malformation rate as documented in women with type 1 diabetes (Bell, Glinianaia et al. 2012).
* In women with pregestational HbA1c < 6.5%, insulin therapy will be initiated either according to capillary maternal blood glucose target values or according to fetal growth assessed by ultrasonography, according to each Diabetes Department habits.

In both groups, care will be standardized as follows:

* Ultrasonography (US) examinations will be performed as usually at 12, 22 and 32 gestational weeks. Additional US will be performed at 25, 28, 35 and 38 gestational weeks, as performed in the several randomized controlled trials that showed that this strategy allows prevention of an increase in the rate of macrosomia in women with GDM (Schaefer-Graf, Kjos et al. 2004). A referent sonographer will be identified in each center to limit the inter-examiner variability. At each US, fetal biometry (with abdominal circumference and fetal weight estimations) and the percentiles according to gestational age will be determined.
* Blood glucose self-monitoring, comprising 6 measures (before and 2 hours after the beginning of each meal), will be registered during a whole week at the end of the three trimesters of pregnancy.
* Women body weight will be measured before pregnancy, at each Diabetology appointment and before delivery.
* Fetal monitoring will be performed according to local routine protocols. Modalities of delivery will be decided as usual care in each obstetrics department. No specific gestational age and modalities of delivery will be recommended for the study.

Group of women with insulin therapy from the beginning of pregnancy :

Treatment will be conducted according to national guidelines for GDM (2010) and consists in:

* Blood glucose self-monitoring before and 2 hrs after each meal, i.e. 6 tests per day. Recommended targets are less than 0.95 g/L before meals and less than 1.20 g/L postprandial.
* Diet counseling with carbohydrate intake divided into three meals and two to three snacks.
* After 7-10 days of glucose monitoring, insulin therapy will be instituted if capillary glucose levels exceed the targets in 20% of all measurements or in 40% of a single time slot. Each caregiver will manage insulin therapy according to local habits (use of long-acting insulin, regular insulin, insulin analogs, continuous subcutaneous insulin infusion by an external pump), and will increase the doses in order to obtain recommended glucose targets. Preliminary data suggest that high insulin doses may be necessary and that normalizing fasting blood glucose may be difficult. Thus, insulin doses will not be further increased in case of the occurrence of repeated hypoglycemia (i.e. 2 mild hypoglycemic episodes in a single slot over one week or one single severe hypoglycemic episode even when blood glucose targets are not achieved).

Insulin treatment will be stopped only in case of fetal restricted growth defined by an estimated fetal weight < 10th percentile, on two consecutive US with at least 3 weeks interval and no other etiology.

Group of women with insulin therapy initiated according to fetal US measurements :

Women will monitor their blood glucose levels before and 2 hours after meals twice a week during the whole pregnancy.

In this group, MODY2 women will not be treated with insulin until delivery, except when:

* the fetal abdominal circumference exceeds ≥ the 75 percentile on one US. This threshold is similar to the one chosen to initiate insulin therapy in several RCTs that showed that this strategy allowed prevention of an increase in the rate of macrosomia in women with GDM (Schaefer-Graf, Kjos et al. 2004, Kjos and Schaefer-Graf 2007).
* or maternal fasting capillary blood glucose is ≥ 1,20 g/L or maternal post-prandial capillary blood glucose is ≥ 2,00 g/L. In the mentioned RCTs, women followed with monthly fetal growth evaluations were not treated with insulin except when fetal abdominal circumference was ≥ 75th percentile, or when their glucose levels exceeded the same safety thresholds. No increase in macrosomia and other pregnancy adverse outcomes was observed using this strategy, as compared to conventional treatment with insulin (Kjos and Schaefer-Graf 2007).

When initiated, insulin therapy will be conducted as described in 11.2, with the same capillary blood glucose targets

-Maternal care Systematic visits in the Diabetes department will be scheduled at 2- 4 weeks intervals. A monthly visit in the Obstetrics department will be scheduled from 22 weeks of gestation.

Routine care, including measurement of weight, height and arterial pressure, as well an urinary testing for proteinuria will be performed at the first appointment and at each following visit.

In case of insulin treatment, the type and dose of insulin will be recorded, as well as the frequency of mild or severe hypoglycemia.

Women with pre-gestational HbA1c > 6.5% will be treated with insulin from the pregnancy planning period or from the beginning of the pregnancy as described in part 6.2.1 and all data concerning these pregnancies will be registered.

* Quality of life Three self-questionnaires, already used in randomized studies of GDM treatment (Crowther, Hiller et al. 2005), will be proposed to all women at the first appointment and at three months post partum.
* Maternal health status will be assessed by means of the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36), which assesses eight aspects of health status: general and mental health, physical and social functioning, physical and emotional role, pain, and vitality. Scores on each scale can range from 0 (worst) to 100 (best).
* Maternal anxiety will be assessed with the use of the short form of the Spielberger State-Trait Anxiety Inventory, a self-rating scale consisting of 6 items (scores below 15 are considered normal).

The presence of a maternal depression will be reflected by a score of more than 12 on the Edinburgh Postnatal Depression Scale at three months post partum.

-Anthropometrics and biological measures in neonates

Anthropometrics parameters will be recorded the first day of life for each neonate:

* Weight to determine "large for gestational age" defined as birth weight above the 90th percentile and "small for gestational age" defined as birth weight below the 10th percentile on sex-specific neonatal growth standards published by the AUDIPOG group (Mamelle et al, 1996)
* Skin fold between 1st and 3rd day of life (bicipital, tricipital, scapular, iliac) for departments experienced in this type of measurement.

Capillary blood glucose test will be collected 3 hours before the first feeding to look for hypoglycaemia. After the second feeding, blood glucose tests will be repeated every 6 hours if > 2.5 mmol/L. If blood glucose is normal during 24 hours and feeding is also normal, neonate glucose monitoring will be stopped.

Infants will be categorized as having clinical neonatal hypoglycaemia if there are symptoms and/or treatment with a glucose infusion or a glucose value ≤ 2 mmol/L.

C-peptide will be measured on cord blood. Hyperinsulinemia is defined by a C-peptide level above the 90th percentile of a neonate reference population. Samples will be centralized in a single laboratory for determination of the C-peptide level.

Neonatal leptin will be measured on cord blood as a biological marker of infant adiposity. Leptin is specifically produced by adipose tissue and placenta, and maternal leptin does not cross the placenta. Fetal leptin reflects the amount of adipose tissue, and its production could be regulated by insulin (Hauguel-de Mouzon, Lepercq et al. 2006).

-GCK genotyping In order to analyze the effect of the maternal treatment according to the fetal genotype, a targeted sequencing of the maternal GCK mutation will be performed on DNA extracted from blood cord sample. The mother (and her partner) will sign an informed written consent for the genetic testing of their baby.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with a GCK mutation before pregnancy
* Aged ≥ 18 years old
* Pre-gestational BMI < 30kg/m²
* Term of pregnancy < 14 WG , if delay overdue, to be validated by investigators
* Written informed consent

Exclusion Criteria:

* Twin pregnancy
* Not able to understand and sign written informed consent
* Not affiliated to the French Social Security

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Birth weight for gestational age | at birth
  this end point will sustain two derived criteria: birth weight for gestational age as a quantitative criterion and birth weight considered as small (below the 10th percentile), normal, or large (above the 90th percentile).

SECONDARY OUTCOMES:
Number of neonatal hypoglycaemia | at birth
  defined as the presence of symptoms and/or the need for treatment with a glucose infusion, and/or a plasma or capillary glucose value ≤ 2 mmol/L within the first 24 hrs
Number of hyperinsulinemia | at birth
  defined by a C-peptide level >90th
Neonatal leptin level | at birth
Number of fetal and neonatal complications | at birth
  Major and minor complications, stillbirth, shoulder dystocia, birth trauma, admission to neonatal intensive care unit, jaundice, respiratory distress syndrome, 5-min Apgar score <7, Cord blood glucose pH<7.2 mmol/L.
Composite obstetrical outcome | at birth
  Gestational age at delivery, mode of delivery, elective cesarean delivery, emergency cesarean delivery, labor induction
Mean blood glucose levels | before and 2 hours post prandial over one week, before pregnancy
Mean blood glucose levels | before and 2 hours post prandial over one week, at weeks 14-16 of pregnancy
Mean blood glucose levels | before and 2 hours post prandial over one week, at weeks 25-27 of pregnancy
Mean blood glucose levels | before and 2 hours post prandial over one week, at weeks 36-38 of pregnancy
Post-prandial hyperglycaemic peak (level and delay) | at 22 weeks of pregnancy
Post-prandial hyperglycaemic peak (level and delay) | at 32 weeks of pregnancy
HbA1c level | pre-gestational and monthly during pregnancy
  according to the HPLC method
Fructosamine level | monthly during pregnancy
Number of women requiring insulin treatment | at 38 weeks of pregnancy
Term of insulin therapy | at 38 weeks of pregnancy
  in case of insulin therapy
Type of insulin | at 38 weeks of pregnancy
  in case of insulin therapy
Number of injections | at 38 weeks of pregnancy
  in case of insulin therapy
Number of units/kg.day of insulin | over one week at weeks 14/16, 25/27 and 36/38
  in case of insulin therapy
Weight gain during pregnancy | at 38 weeks of pregnancy
Number of pregnancy induced hypertension | at delivery
  to evaluate maternal complications
Number of preeclampsia | at delivery
  to evaluate maternal complications
Number of medical appointments | at delivery
  to evaluate maternal complications
Duration of hospital stay | at delivery
  to evaluate maternal complications
depression (Edinburgh Postnatal Depression Scale. | at delivery
  to evaluate maternal complications
Quality of Life (SF-36 questionary) | at delivery
  to evaluate maternal complications
Anxiety score (short form of the Spielberger State - Trait Anxiety Inventory | at delivery
  to evaluate maternal complications

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bellanné-Chantelot, PharmaD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- La Pitié Salpêtrière Hospital, Paris, France

REFERENCES:
- [Derived] Ciangura C, Seco A, Saint-Martin C, Ancel PY, Bouvet D, Jacqueminet S, Hartemann A, Lepercq J, Nizard J, Timsit J, Bellanne-Chantelot C; Monogenic Diabetes Study Group of the Societe Francophone du Diabete. Pregnancy and neonatal outcomes in women with GCK-MODY: an observational study based on standardised insulin modalities. Diabetologia. 2025 May;68(5):981-992. doi: 10.1007/s00125-025-06363-0. Epub 2025 Feb 19. PMID 39971752